CLINICAL TRIAL: NCT04095975
Title: Effectiveness of Prescription vs. Non-prescription Urinary Alkalinizing Agents on Kidney Stone Risk
Brief Title: Effectiveness of Urinary Alkalinizing Agents on Kidney Stone Risk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0621; A539800 (Other: UW Madison); SMPH/UROLOGY/UROLOGY (Other: UW Madison); Protocol Version 9/9/2020 (Other: UW Madison)
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baking Soda (Active Comparator): Subjects randomized to baking soda will be provided instructions for using baking soda to provide 40 mEq alkali, to be accomplished by dissolving ¼ teaspoon baking soda in water or other beverage (any amount) in the morning on an empty stomach and ½ teaspoon baking soda in water or other beverage again at bedtime, also on an empty stomach.
  Interventions: Dietary Supplement: Baking Soda
- LithoLyte (Active Comparator): Subjects randomized to LithoLyte® will be provided 40 mEq of alkali in the form of LithoLyte® and advised to take 20 mEq twice daily according to package instructions, once in morning and once at bedtime; no requirements about proximity to meals are necessary.
  Interventions: Dietary Supplement: LithoLyte

INTERVENTIONS:
Dietary Supplement: Baking Soda — Standard baking soda that can be bought from stores.
  Arms: Baking Soda
Dietary Supplement: LithoLyte — LithoLyte is considered a medical food and consists of: potassium citrate, magnesium citrate, sodium bicarbonate, and erythritol.
  Arms: LithoLyte

SUMMARY:
Randomized treatment trial of baking soda or LithoLyte to determine if baking soda and Litholyte are effective in raising 24 hour urine citrate and pH.

DETAILED DESCRIPTION:
Participants will not be required to attend any study visits outside of normal clinical encounters. Participants enrolled in the study will be randomized to treatment upon enrollment. Blocked randomization will be conducted, utilizing sex (M/F) and recurrent stone former (Y/N) as algorithm variables.

Participants randomized to LithoLyte® will be provided 40 mEq of alkali in the form of LithoLyte® and advised to take 20 mEq twice daily according to package instructions, once in morning and once at bedtime; no requirements about proximity to meals are necessary.

Participants randomized to baking soda will be provided instructions for using baking soda to provide 40 mEq alkali, to be accomplished by dissolving ¼ teaspoon baking soda in water or other beverage (any amount) in the morning on an empty stomach and ½ teaspoon baking soda in water or other beverage again at bedtime, also on an empty stomach.

The 24-hour urine results that are available upon enrollment will be used for pre-intervention values. The 24-hour results from each participant's followup collection will be used for post-intervention values. Thus, no extra encounters are required for participation in the study. Additionally, no extra tests are required for participation in the study as participants would normally complete a post-treatment 24-hour urine collection anyway. Participants will be screened for eligibility, i.e., by pre-clinic review of schedules and 24-hour urine results. Only those meeting inclusion criteria will be invited to participate and enrolled, provided that informed consent is provided by signing the signature page of the consent/authorization form. The treatment/intervention period is up to 90 days (approximately 3 months). However, it should be noted that, as these are clinical interventions that would be prescribed or recommended anyway, it is expected that participants will continue treatment indefinitely and under supervision of urology and/or Metabolic Stone Clinic providers. If the participant has failed the randomized therapy they are assigned to, they will be clinically assigned a different treatment option and continue to be followed up in routine fashion.

Participants will also be asked to complete a medication questionnaire and log, as well as the Wisconsin Stone Quality of Life (WISQOL) questionnaire. All study procedures are considered standard of care, except for: randomization into treatment and the medication questionnaire and log.

Protocol Amendment Approved 11/16/2020 removed the UrocitK study arm; the investigators faced challenges recruiting participants during the COVID-19 pandemic and the possibility of being randomized into a prescription drug arm was causing many potential participants to choose not to participate.

ELIGIBILITY:
Inclusion Criteria:

* Must be suitable for the study per clinical judgement of study team members
* Patient in the UW Health University Hospital Urology Clinic or the Metabolic Stone Clinic
* Had at least one kidney stone event
* Greater than or equal to 18 years of age
* 24 hour urine citrate is less than 420 mg and/or urine pH is less than 5.9
* Urinary alkalinization is deemed by provider as a necessary therapeutic goal for the subject and may be achieved by any of the three therapies under examination
* Subject is willing to provide consent and to be randomized into a treatment

Exclusion Criteria:

* Subject is deemed unsuitable for urinary alkalinizing therapy by study staff
* Subject is already on a urinary alkalinizing agent
* Subject is on acetazolamide
* Subject reports sensitivity to sugar alcohols
* Subject is under 18 years of age
* Subject has not completed a 24 hour urine collection within 6 months
* Subject is pregnant or breastfeeding
* Subject is unable or unwilling to provide consent
* Subject is unable or unwilling to be randomized
* Subject reports they are unwilling or unable to use measuring device required in the baking soda arm of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Change in 24 hour urine citrate | Pre and 24 hour post intervention (up to 90 days)
  Pre-to-post intervention change in 24-hour urine citrate will be measured
  Reference range of Urine Citrate:
  18 years and older: 320-1240 mg/d
  1 year and older: greater than or equal to 150 mg/g.
Change in 24 hour urine pH | Pre and 24 hour post intervention (up to 90 days)
  Pre-to-post intervention change in 24-hour urine pH will be measured
  Reference range of Urine pH:
  Age 0 days and up: 5.0-8.0

SECONDARY OUTCOMES:
Post-intervention 24-hour urine calcium | Enrollment and follow up visit (approximately 90 days)
  Urine calcium levels will be measured post intervention.
  Reference range of Urine Calcium:
  0-17 years: up to 6.0 mg/kg/24 hours 18 years and up: 100-300 mg/24 hours
24 hour urine calcium | Enrollment and follow up visit (approximately 90 days)
  Reference range of urine calcium:
  0-12 years: 7-31 mg/d Male 13 years and older: 16-49 mg/d Female 13 years and older: 13-40 mg/d
Post interventional 24 hour urine supersaturation indices for calcium oxalate | Enrollment and follow up visit (approximately 90 days)
  Supersaturation means there are too many salts and not enough fluids in the urine. It's the driving force behind stone formation. Post interventional 24 hour urine supersaturation indices for calcium oxalate will be measured.
  Reference range:
  0-12 years: 7-31 mg/d Male 13 years and older: 16-49 mg/d Female 13 years and older: 13-40 mg/d
Post interventional 24 hour urine supersaturation indices for calcium phosphatase | Enrollment and follow up visit (approximately 90 days)
  Supersaturation means there are too many salts and not enough fluids in the urine. It's the driving force behind stone formation. Post interventional 24 hour urine supersaturation indices for calcium phosphatase will be measured.
  Reference range:
  Age 18 years and up: 0.4-1.3 g/24 hour
Cost of Treatment as measured by USD spent on the interventional drug | End of study (approximately 90 days)
  Cost of baking soda versus LithoLyte.
Patient acceptability | End of study (approximately 90 days)
  Wisconsin Stone-QOL: answers range from a scale of 1-5, or yes/no
  Study Questionnaire: free text responses, or no/yes/I am no longer taking it

CONTACTS AND LOCATIONS:
Overall Officials: Kristina L Penniston, PhD, RDN, FAND, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No